CLINICAL TRIAL: NCT07287007
Title: Evaluating the Hemodynamic Performance of the VenAir Sequential Compression System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wellell Inc. Taiwan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: EC1140707-F
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: No Condition, Healthy Individuals; No Conditions, Aged 20-64
Keywords: Intermittent pneumatic compression; Hemodynamics; Venous thromboembolism prophylaxis

STUDY DESIGN:
Intervention Model Description: This study uses a randomized crossover design in which each participant will be tested with two devices (VenAir and SCD700). The same participant will use both devices, allowing each participant to serve as their own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VenAir (Experimental): The VenAir and its garments (thigh, calf, foot) will be tested in a randomized testing order.
  Interventions: Device: VenAir
- SCD700 (Active Comparator): The SCD700 and its garments (thigh, calf, foot) will be tested in a randomized testing order.
  Interventions: Device: SCD700

INTERVENTIONS:
Device: VenAir — VenAir is an intermittent pneumatic compression (IPC) device intended to help prevent venous thromboembolism (VTE), including deep vein thrombosis (DVT) and pulmonary embolism (PE). In this study, VenAir is applied to the participant's lower limb under standard operating settings, and hemodynamic performance is measured for comparison with SCD700.
  Arms: VenAir
Device: SCD700 — SCD700 is a commercially available intermittent pneumatic compression (IPC) device used to prevent venous thromboembolism (VTE), including deep vein thrombosis (DVT) and pulmonary embolism (PE). In this study, SCD700 is applied to the participant's lower limb under standard operating settings, and hemodynamic performance is measured to compare with VenAir.
  Arms: SCD700

SUMMARY:
The goal of this clinical trial is to learn an Intermittent Pneumatic Compression Device (IPCD), VenAir, effectiveness in healthy adults. The main questions this research aims to answer are:

1. The hemodynamic performance of VenAir paired with the thigh garments, calf garments, and foot garments is not inferior to that of SCD700 paired with the corresponding garments.
2. The hemodynamic performance of VenAir paired with the thigh garments, calf garments, and foot garments is not inferior to that of SCD700 paired with the thigh garment.

Researchers will compare VenAir and the SCD700 to see if the hemodynamic performance of VenAir is as well as or not worse than the SCD700.

Participants will lie down and rest for approximately 30 minutes to stabilize their heart rate. The researcher will then use ultrasound to measure the participant's blood flow while they wear different leg garments (one at a time) and also when no garment is worn.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Aged 20-64 years
* Leg circumference within the size range of the SCD700 and VenAir garments

Exclusion Criteria:

* Cardiovascular-related diseases (mild atherosclerosis, other ischemic vascular diseases, congestive heart failure, etc.)
* Previous suspicion of deep vein thrombosis, pulmonary embolism, or phlebitis
* History of stroke
* History of varicose vein surgery
* Hypertension
* Diabetes
* Dermatitis, gangrene, or severe wounds
* Massive edema of legs
* Pregnancy
* Pulmonary edema

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-10-05 (Estimated); Study Completion 2026-10-05 (Estimated)

PRIMARY OUTCOMES:
Peak Velocity of Blood Flow Increasement | During and immediately after device application
  The peak velocity increasement is measured to understand the degree of change in peak blood flow velocity with and without using the IPC device. Baseline peak velocity is calculated by averaging the two highest peaks over a 16-second period without the device. Intervention peak velocity is obtained by averaging the peak velocities over four compression cycles while wearing the IPC device.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Yung Chang, Principal Investigator — Wellell Inc.
Locations (1):
- Wellell Inc., New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muhe E. Intermittent sequential high-pressure compression of the leg. A new method of preventing deep vein thrombosis. Am J Surg. 1984 Jun;147(6):781-5. doi: 10.1016/0002-9610(84)90200-9. PMID 6731693
- [Background] Kamm R, Butcher R, Froelich J, Johnson M, Salzman E, Shapiro A, Strauss HW. Optimisation of indices of external pneumatic compression for prophylaxis against deep vein thrombosis: radionuclide gated imaging studies. Cardiovasc Res. 1986 Aug;20(8):588-96. doi: 10.1093/cvr/20.8.588. PMID 3791348
- [Background] Labropoulos N, Giuliano KK, Tafur AJ, Caprini JA. Comparison of a nonpneumatic device to four currently available intermittent pneumatic compression devices on common femoral blood flow dynamics. J Vasc Surg Venous Lymphat Disord. 2021 Sep;9(5):1241-1247. doi: 10.1016/j.jvsv.2021.01.008. Epub 2021 Feb 1. PMID 33540132
- [Background] 1. Virchow RLK. Die Verstopfung den Lungenarterie und ihre Folgen. Beitr Exper Path Physiol. 1846;2(1). 2. Pavon JM, Adam SS, Razouki ZA, et al. Effectiveness of Intermittent Pneumatic Compression Devices for Venous Thromboembolism Prophylaxis in High-Risk Surgical Patients: A Systematic Review. J Arthroplasty. 2016;31(2):524-532. doi:10.1016/j.arth.2015.09.043 3. Anderson DR, Morgano GP, Bennett C, et al. American Society of Hematology 2019 guidelines for management of venous thromboembolism: prevention of venous thromboembolism in surgical hospitalized patients. Blood Advances. 2019;3(23):3898-3944. doi:10.1182/bloodadvances.2019000975 4. Reitsma PH, Versteeg HH, Middeldorp S. Mechanistic View of Risk Factors for Venous Thromboembolism. ATVB. 2012;32(3):563-568. doi:10.1161/ATVBAHA.111.242818 5. Sadaghianloo N, Dardik A. The efficacy of intermittent pneumatic compression in the prevention of lower extremity deep venous thrombosis. Journal of Vascular Surgery: Venous and Lymphatic Disorders. 2016;4(2):248-256. doi:10.1016/j.jvsv.2015.07.006 6. Kakkos SK, Szendro G, Griffin M, Daskalopoulou SS, Nicolaides AN. The efficacy of the new SCD Response Compression System in the prevention of venous stasis. Journal of Vascular Surgery. 2000;32(5):932-940. doi:10.1067/mva.2000.110358 7. Kakkos SK, Szendro G, Griffin M, Sabetai MM, Nicolaides AN. Improved hemodynamic effectiveness and associated clinical correlations of a new intermittent pneumatic compression system in patients with chronic venous insufficiency. Journal of Vascular Surgery. 2001;34(5):915-922. doi:10.1067/mva.2001.118822 8. Morris RJ. Intermittent pneumatic compression - systems and applications. J Med Eng Technol. 2008;32(3):179-188. doi:10.1080/03091900601015147
- [Background] Kakkos SK, Szendro G, Griffin M, Sabetai MM, Nicolaides AN. Improved hemodynamic effectiveness and associated clinical correlations of a new intermittent pneumatic compression system in patients with chronic venous insufficiency. J Vasc Surg. 2001 Nov;34(5):915-22. doi: 10.1067/mva.2001.118822. PMID 11700495
- [Background] Kakkos SK, Szendro G, Griffin M, Daskalopoulou SS, Nicolaides AN. The efficacy of the new SCD response compression system in the prevention of venous stasis. J Vasc Surg. 2000 Nov;32(5):932-40. doi: 10.1067/mva.2000.110358. PMID 11054225
- [Background] Sadaghianloo N, Dardik A. The efficacy of intermittent pneumatic compression in the prevention of lower extremity deep venous thrombosis. J Vasc Surg Venous Lymphat Disord. 2016 Apr;4(2):248-56. doi: 10.1016/j.jvsv.2015.07.006. Epub 2015 Sep 15. PMID 26993875
- [Background] Reitsma PH, Versteeg HH, Middeldorp S. Mechanistic view of risk factors for venous thromboembolism. Arterioscler Thromb Vasc Biol. 2012 Mar;32(3):563-8. doi: 10.1161/ATVBAHA.111.242818. PMID 22345594
- [Background] Anderson DR, Morgano GP, Bennett C, Dentali F, Francis CW, Garcia DA, Kahn SR, Rahman M, Rajasekhar A, Rogers FB, Smythe MA, Tikkinen KAO, Yates AJ, Baldeh T, Balduzzi S, Brozek JL, Ikobaltzeta IE, Johal H, Neumann I, Wiercioch W, Yepes-Nunez JJ, Schunemann HJ, Dahm P. American Society of Hematology 2019 guidelines for management of venous thromboembolism: prevention of venous thromboembolism in surgical hospitalized patients. Blood Adv. 2019 Dec 10;3(23):3898-3944. doi: 10.1182/bloodadvances.2019000975. PMID 31794602
- [Background] Pavon JM, Adam SS, Razouki ZA, McDuffie JR, Lachiewicz PF, Kosinski AS, Beadles CA, Ortel TL, Nagi A, Williams JW Jr. Effectiveness of Intermittent Pneumatic Compression Devices for Venous Thromboembolism Prophylaxis in High-Risk Surgical Patients: A Systematic Review. J Arthroplasty. 2016 Feb;31(2):524-32. doi: 10.1016/j.arth.2015.09.043. Epub 2015 Oct 29. PMID 26525487
- [Background] Virchow RLK. Die Verstopfung den Lungenarterie und ihre Folgen. Beitr Exper Path Physiol. 1846;2(1).